CLINICAL TRIAL: NCT01496339
Title: Phase 1/2 Clinical Study of MenSCs Infusion in Type 1 Diabetes
Brief Title: Human Menstrual Blood-derived Mesenchymal Stem Cells Transplantation in Treating Type 1 Diabetic Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: S-Evans Biosciences Co., Ltd. (Industry)
Collaborators: Zhejiang University (Other); Wenzhou Medical University (Other); Zhenjiang First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEB-1213-T1DM
Record Dates: First submitted 2011-12-18; First posted 2011-12-21 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional therapy control (Active Comparator)
  Interventions: Drug: exogenous indulin injection daily
- Stem cell infusion (Experimental)
  Interventions: Biological: MenSCs transplantation

INTERVENTIONS:
Biological: MenSCs transplantation — 1×10^6/kg MenSCs are infused through pancreatic artery or intravenous infusion once a week by the 4 consecutive therapies.
  Arms: Stem cell infusion
Drug: exogenous indulin injection daily — traditional therapy, such as insulin injection daily, monitoring random and postprandial blood glucose.
  Arms: Traditional therapy control

SUMMARY:
The purpose of this study is to investigate whether the treatment of human menstrual blood-derived mesenchymal stem cells which would be applied to diabetes patients is safe and effective.

DETAILED DESCRIPTION:
Diabetes mellitus is chronic metabolic diease caused by absent or rejection insulin from pancreatic b cells.The traditional treatment strategies for diabetes are daily injections with insulin and transplantation of islets from cadaver. However, daily injuection is very inconvenient and there is a shortage of organs and life long immunosuppression. Therefore, such therapy can be offered to a very limited number of patients only. MSC-based therapeutic intervention has become an emerging strategy for the replacement of injured tissues. MSCs also have been noted to possess immunomodulatory effects in vivo. Thus, their potential for clinical use as a cell-based therapy should be focused and observation.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients at the age of 18 to 75.
* agreement to receive written informed consent.
* voluntary submission to the procedures of the study protocol.
* clinical diagnosis is classified to type 1 diabetes(T1DM).
* T1DM duration ≥ 1 and ≤ 20 years from the time of enrollment.

Exclusion Criteria:

* renal dysfunction, eye disease or other organ disease.
* cardiovascular disease, existing congestive cardiac failure on physical exam and/or acute coronary syndrome in past 6 months.
* pregnancy
* mental disorders
* hepatitis C, HIV, RPR,active tuberculosis or blood diseases
* any malignancy
* any other severe diseases that could potentially influence the infusion results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Glycosylated hemoglobin (HbA1c) | 1 year

SECONDARY OUTCOMES:
The acute reaction and severity of adverse events related to the stem cell infusion procedure | 2 years
Number of severe and documented hypoglycemic events | 2 years
C-peptide release test | 3 months
The reduction in fasting blood glucose (FBG) | 1 year
The increase in basal C-peptide | 1 year
The postprandial blood glucose | 1 year
The random glucose level | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Charile Xiang, Professor, Principal Investigator — S-Evans Biosicences Co.,Ltd
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China